CLINICAL TRIAL: NCT05958875
Title: A Randomised, Controlled Trial to Investigate the Effect of a Six Week Intensified Pharmacological Treatment for Schizophrenia Compared to Treatment as Usual in Subjects Who Had a First-time Treatment Failure on Their First-line Treatment.
Brief Title: The Effect of a Six Week Intensified Pharmacological Treatment for Schizophrenia Compared to Treatment as Usual in Subjects Who Had a First-time Treatment Failure on Their First-line Treatment.
Acronym: INTENSIFY SZ
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Inge Winter (Other)
Collaborators: Universität Münster (Other)
Responsible Party: Sponsor-Investigator, Dr. Inge Winter, Principal Investigator, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-506602-39-00 (EU CT#)
Record Dates: First submitted 2023-06-30; First posted 2023-07-25 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia and Related Disorders; Early Treatment-Resistance
Keywords: Schizophrenia; Schizoaffective disorder; Schizophreniform disorder; Clozapine; Treatment as usual; Early treatment-Resistance
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Clozapine; Therapeutics

STUDY DESIGN:
Intervention Model Description: Parallel randomization to the 2 arms, treatment as usual (TAU) or early-intensified pharmacological treatment (EIPT).
Who Masked: Outcomes Assessor
Masking Description: Open label, except for the assessors of the primary outcome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schizophrenia early intensified treatment (EIPT): Switch to clozapine (Experimental): Subject with schizophrenia, randomized to EIPT: Switch to clozapine. Brand, dosage, frequency and duration up to the investigator's discretion
  Interventions: Drug: Clozapine
- Schizophrenia treatment as usual (TAU): second-line antispychotic (Active Comparator): Subject with schizophrenia or related disorder randomized to TAU: switch to second-line antispychotic. Compound, brand, dosage, frequency and duration up to the investigator's discretion (in accordance with SmPC)
  Interventions: Drug: Second-line Antipsychotics (treatment as usual)

INTERVENTIONS:
Drug: Clozapine — Participants are randomized to clozapine or second-line antipsychotics. When randomised to clozapine, they will receive clozapine for six weeks.
  Other Names: ATC code: N05AH02
  Arms: Schizophrenia early intensified treatment (EIPT): Switch to clozapine
Drug: Second-line Antipsychotics (treatment as usual) — Participants are randomized to clozapine or second-line antipsychotics. When randomized to second-line antipsychotics, this means participants will receive treatment as usual. The physician has the choice to administer any second-line antipsychotic. More specification is not possible, as this is a choice the physician makes with the participant based on the characteristic and preference of the participant (in line with standard clinical practice).
  Arms: Schizophrenia treatment as usual (TAU): second-line antispychotic

SUMMARY:
Schizophrenia (SZ) affects approximately 4.5 million people across the European Union (EU) and is associated with annual healthcare and societal costs of 29 billion Euros. The impact on the daily life of patients is huge, ranging from frequent relapses and hospitalisations, the inability to maintain a job or continue scholing, to a low quality of life, impaired cognitive functioning, suicidal ideation and an increase morbidity rate, next to the large burden for carers 1. When diagnosed with schizophrenia or related disorder, patients are commonly prescribed antipsychotics. One-third of the schizophrenia patients are regarded treatment-resistant (TR), meaning that at least two antipsychotic trials have failed. Typically, clozapine is prescribed for TR patients, which is effective for approximately 40% of patients. Clozapine is among the most effective treatments, with the lowest all-cause mortality. Although it is among the most effective antipsychotics, it is generally not used earlier in the illness course due to a small risk of severe neutropenia/agranulocytosis, which is why patients treated with clozapine are intensely monitored. However, this small risk outweighs the burden of not receiving an effective treatment.

Since clozapine is among the most effective treatments, this leads to the research question whether earlier initiation of third-line treatment ('early intensified' pharmacological treatment; EIPT) would be more beneficial than the current second-line treatments (treatment as usual; TAU). If this is indeed the case, this could lead to the prevention of unnecessary trials of ineffective treatments, hospitalisations, and recommendations for adaptations of worldwide guidelines as well as a reduction of healthcare and societal costs The INTENSIFY-Schizophrenia trial is part of the larger Horizon 2021 project Psych-STRATA, with the central goal of paving the way for a shift towards a treatment decision-making process tailored for the individual at risk for treatment resistance. To that end, the inestigators aim to establish evidence-based criteria to make decisions of early intense treatment in individuals at risk for treatment resistance across the major psychiatric disorders of schizophrenia, bipolar disorder and major depression. The current protocol focuses on the sample of schizophrenia patients.

DETAILED DESCRIPTION:
Rationale Schizophrenia (SZ) affects approximately 4.5 million people across the European Union (EU) and is associated with annual healthcare and societal costs of 29 billion Euros. The impact on the daily life of patients is huge, ranging from frequent relapses and hospitalisations, the inability to maintain a job or continue scholing, to a low quality of life, impaired cognitive functioning, suicidal ideation and an increase morbidity rate, next to the large burden for carers. When diagnosed with schizophrenia or related disorder, patients are commonly prescribed antipsychotics. One-third of the schizophrenia patients are regarded treatment-resistant (TR), meaning that at least two antipsychotic trials have failed. Typically, clozapine is prescribed for TR patients, which is effective for approximately 40% of patients. Clozapine is among the most effective treatments, with the lowest all-cause mortality. Although it is among the most effective antipsychotics, it is generally not used earlier in the illness course due to a small risk of severe neutropenia/agranulocytosis, which is why patients treated with clozapine are intensely monitored. However, this small risk outweighs the burden of not receiving an effective treatment.

Since clozapine is among the most effective treatments, this leads to the research question whether earlier initiation of third-line treatment ('early intensified' pharmacological treatment; EIPT) would be more beneficial than the current second-line treatments (treatment as usual; TAU). If this is indeed the case, this could lead to the prevention of unnecessary trials of ineffective treatments, hospitalisations, and recommendations for adaptations of worldwide guidelines as well as a reduction of healthcare and societal costs The INTENSIFY-Schizophrenia trial is part of the larger Horizon 2021 project Psych-STRATA, with the central goal of paving the way for a shift towards a treatment decision-making process tailored for the individual at risk for treatment resistance. To that end, the investigators aim to establish evidence-based criteria to make decisions of early intense treatment in individuals at risk for treatment resistance across the major psychiatric disorders of schizophrenia, bipolar disorder and major depression. The current protocol focuses on the sample of schizophrenia patients.

Objective The primary objective is to compare the treatment response, expressed as mean change in symptom severity as measured through the Positive And Negative Syndrome Scale (PANSS) under an early-intensified pharmacological treatment to that under treatment as usual, in subjects who had a first-time treatment failure on their first-line treatment for schizophrenia, schizoaffective or schizophreniform disorder.

Main trial endpoints Mean change in symptom severity total score from baseline (visit 2) to end of treatment (visit 4) between the two treatment arms (EIPT vs. TAU). This is measured using PANSS.

Secondary trial objectives

1. To compare changes in PANSS subscale scores (positive, negative and general) between the two treatment arms.
2. To compare changes in severity and improvement in global functioning assessed by the Clinical Global Impression Scale (CGI) between the two treatment arms.
3. To compare changes in the levels of depression and anxiety between treatment arms.
4. To compare changes in quality of life and functioning measures between treatment arms.
5. To compare changes in cognitive performance between treatment arms.
6. To compare the proportion of participants (EIPT vs. TAU) that is in symptomatic remission at visit 4.
7. To compare presence of adverse events (related and unrelated to treatment) between treatment arms.
8. To compare use of concomitant medication between treatment arms.
9. To compare premature treatment discontinuation (timing and reason) between treatment arms.
10. To compare changes in suicidal ideation between treatment arms.

Trial design The clinical study is an international, multicenter controlled, randomised, open label trial (with blinded raters), with a treatment duration of six weeks.

Trial population The aim is to recruit 418 subjects with schizophrenia, schizoaffective disorder or schizophreniform disorder. Male and female subjects, in- and out-patients, within the age range of 18 to 70 years old are eligible for participation. The main exclusion criteria are defined to protect the wellbeing of subjects, e.g. being pregnant or breastfeeding, subjects with previous failure on clozapine, meeting any contraindications, or participants with a known intolerance to clozapine.

Interventions Subjects are randomised to treatment as usual (second-line treatment) or to the early-intensified pharmacological treatment (third-line treatment; clozapine).

Ethical considerations relating to the clinical trial including the expected benefit to the individual subject or group of subjects represented by the trial subjects as well as the nature and extent of burden and risks All medications studied in the current trial are widely used (alone or in combination) in clinical practice and side effect profiles are well established. In the current study, clinical practice is mimicked as much as possible to maximize generalizability and for feasibility purposes. To this end, Summaries of Product Characteristics (SmPCs) are followed with regards to contraindications (implemented as exclusion criterion), safety measures and prohibited comedications. Site visits and assessments are kept to a minimum to keep subject burden at an acceptable level, while meeting the objectives of the study. Blood samples for biomarker analyses are only collected when subjects provide consent; safety measures are performed as part of clinical routine.

Overall, the risks are similar to daily clinical practice; the only difference relative to clinical practice is the application of early-intensified pharmacological treatment earlier in the illness. Still, these intense treatment options are also commonly prescribed by clinicians. There are no indications in existing literature or clinical practice that the earlier introduction of these medications poses a safety risk when used in an earlier illness phase than indicated in the SmPC.

A benefit of the study is that if it indeed turns out that the clozapine is associated with more symptom improvement compared to treatment as usual, future patients have to go through less trial and error, which results in a reduced burden (higher quality of life, less unemployment, less hospitalisations) for patients and carers as well as lower societal and healthcare costs.

IMPORTANT: the study was submitted to the European authorities before (see NCT05603104) and they requested to split this study into 3 studies (1 for each diagnostic category). We have done this and created 3 new ClinicalTrials.gov studies as well, from which this is one for schizophrenia. For the BD study it is NCT05973786 and for MDD NCT05973851. The site in the UK (London) followed the advice and will submit 3 separate protocols and are therefore included in the current record. However, Israel already submitted this as one protocol. Therefore, we keep the old clinicaltrials.gov number for Israel (NCT05603104).

ELIGIBILITY:
Inclusion Criteria:

1. In- or out patients, at least 18 years of age up until 70.
2. Being willing and able to provide written informed consent. Having a legal guardian to cosign is allowed. Informed consent will be signed at visit 1, before any study procedure.
3. Female subjects of child bearing potential must use effective contraception during the trial as per the requirements of the applicable SmPCs and should have a negative pregnancy test at visit 1 or 2 (before randomisation; section 8.2).
4. Meeting diagnostic criteria for a primary diagnosis of schizophrenia, schizoaffective disorder, or schizophreniform disorder, according to DSM-5. The primary diagnosis will be confirmed by the Mini International Neuropsychiatric Interview (MINI v7.0.2).
5. Subject experiences a treatment failure due to lack of efficacy in the current episode, as confirmed by a CGI-I ≥3; preferably this treatment is a first-line pharmacotherapeutic agent for the primary DSM-5 diagnosis, and was prescribed for at least 4 weeks within an effective dose range as specified in the Summary of Product Characteristics (SmPCs). However, other lines of treatment are accepted as well.
6. Subject and clinician intend to change pharmacotherapeutic treatment.
7. A minimum symptom severity threshold needs to be present (moderate level; see below) and subject needs to experience functional impairment.

   * The minimum symptom severity threshold is at least 2 PANSS positive or negative items with a score of 4, or at least one PANSS positive or negative item with a score of 5.
   * Functional impairment is defined as a score of 5 or higher on any of the three scales of the Sheehan Disability Scale (SDS).

Exclusion criteria:

1. Being pregnant or breastfeeding.
2. Subject has used clozapine in the past.
3. Subject has a known intolerance to clozapine or to all TAU medication options.
4. Meeting any of the contraindications of clozapine or to all TAU medication options, as specified within the applicable SmPC.
5. Subject has participated in another clinical trial in which the subject received an experimental or investigational drug or agent within 30 days before visit 1.
6. Subject experiences any other significant disease or disorder which, in the opinion of the investigator, may either put the subjects at risk because of participation in the trial, or may influence the result of the trial, or the subject's ability to participate in the trial.
7. Subjects with active suicidal ideation with some intent to act, without specific plan ("Yes" to question 4 of the Columbia-Suicide Severity Rating Scale (C-SSRS)) or active suicidal ideation with specific plan and intent ("Yes" to question 5 of the C-SSRS), followed by an assessment by the treating clinician who determines it is not safe for the subject to participate in the study
8. Subject meets criteria for current substance use disorder, as confirmed by the Mini International Neuropsychiatric Interview (MINI v7.0.2). Nicotine dependency is allowed, as well as mild and moderate alcohol and/or cannabis use disorder (as defined by MINI v7.0.2). Severe alcohol and/or cannabis use disorder are not allowed.
9. Subjects have not been committed to an institution by virtue of an order issued either by the judicial or the administrative authorities.
10. Subjects who meet the modified Andreasen criteria for remission.
11. Subjects that have any clinically significant abnormal values on the local laboratory test (especially ANC/WBC and liver values), electrocardiogram (ECG) or physician examinations.
12. Subjects dependent on the sponsor, investigator or trial site must be excluded from participation in advance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in symptom severity on Positive and Negative Syndrome Scale | 6 weeks
  Change in symptom severity (EIPT vs. TAU) total score from baseline (visit 2) to end of treatment (visit 4). This is measured using the Positive And Negative Syndrome Scale. Minimum score is 30, maimum score 210. A bigger mean change means a better outcome.

SECONDARY OUTCOMES:
Compare symptomatic remission. | 6 weeks
  Comparison of the proportion of participants (EIPT vs. TAU) that is in symptomatic remission at visit 4. Remission is defined as meeting all the Positive and Negative Syndrome Scale modified Andreasen criteria (Low scores (≤3) P1. Delusions; P3. Hallucinatory behavior; P2. Conceptual disorganization; N1. Blunted affect; N4. Passive/apathetic social withdrawal; N6. Lack of spontaneity and flow of conversation; G5. Mannerisms/posturing; G9. Unusual thought content. There is no minimum or maximum score; either a participants meets the criteria or not (dichotomous outcome).
To compare changes in PANSS subscale scores (positive, negative and general) between the two treatment arms. | 6 weeks
  To compare changes in Positive and Negative Syndrome Scale subscale scores (positive (mimumum score 7, maximum score 49), negative (minimum score 7, maximum score 49) and general( (minimum score 16, maximum score 112)) between the two treatment arms over the six-week treatment period (visit 2 versus visit 4). Lower scores mean better outcomes.
Compare changes in the levels of depression and anxiety | 6 weeks
  To compare changes in the levels of depression and anxiety as assessed with the Hospital Anxiety and Depression Scale between the two treatment arms (EIPT/TAU) over the six week treatment period (visit 2 versus visit 4). Lower scores mean less depression and anxiety.
To compare changes in cognitive performance as measured through the Trail Making Test | 6 weeks
  To compare changes in cognitive performance as measured through the Trail Making Test between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4). A lower time to complete the test means better cognitive performance.
To compare changes cognitive performance as measured through the Digit Symbol Substitution Test | 6 weeks
  To compare changes cognitive performance as measured through the Digit Symbol Substitution Test between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4). A higher scores means better cognitive performance.
To compare changes in cognitive performance as measured through the Rey Auditory Verbal Learning Test | 6 weeks
  To compare changes in cognitive performance as measured through the Rey Auditory Verbal Learning Test between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4). Higher scores means better cognitive performance. There are several scores to calculate: RAVLT Immediate score: the sum of scores from 5 first trials (Trials 1 to 5).
  RAVLT Learning score: the score of Trial 5 minus the score of Trial 1. RAVLT Forgetting: the score of Trial 5 minus score of the delayed recall. RAVLT Percent Forgetting score: RAVLT Forgetting divided by the score of Trial 5.
To compare changes in subjective cognitive performance as measured through the Perceived Deficits Questionnaire | 6 weeks
  To compare changes in cognitive performance as measured through the Perceived Deficits Questionnaire between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4). A higher scores means worse subjective cognitive performance.
To compare changes in functioning on the Leuven Afective and Pleasure Scale | 6 weeks
  To compare changes in the functioning measure, Leuven Afective and Pleasure Scale, between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4). A higher scores means worse functioning. Minimum score: 0, Maximum score: 160
To compare changes in functioning on the Sheehan Disability Scale | 6 weeks
  To compare changes in the functioning measure,Sheehan Disability Scale, between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4). A higher scores means worse functioning. Minimum score: 0, maximum score 30.
To compare changes in quality of life measure, Quality of Life Enjoyment and Satisfaction Questionnaire Short Form | 6 weeks
  To compare changes in quality of life measure, Quality of Life Enjoyment and Satisfaction Questionnaire Short Form between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4). A higher scores means better quality of life. Minimum score: 16, maximum score: 80.
To compare changes in quality of life measure, Quality of Life Scale -100, subscale inner tension | 6 weeks
  To compare changes in quality of life measure, Quality of Life Scale -100, subscale inner tension between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4). This is a dichotomous scale (unsatisfactory or satisfactory). More 'satisfatory' answers means higher quality of life.
To compare presence of adverse events (related and unrelated to treatment) between treatment arms. | 6 weeks
  To compare presence of adverse event (related and unrelated) as measured through General Assessment of Side Effects Scale and reported spontaneously between the two treatment arms (EIPT/TAU) over the six week treatment period (visit 2 versus visit 4). Higher scores means more side effects. Minimum score: 0 side effects, maximum score: 38 side effects.
To compare the use of concomitant medication between the two treatment arms. | 6 weeks
  To compare use of concomitant medication between the two treatment arms (EIPT/TAU) over the six week treatment period (visit 2 versus visit 4).
To compare the difference in number of participants (EIPT vs. TAU) that prematurely discontinuate the study treatment. | 6 weeks
  To compare the difference in number of participants (EIPT vs. TAU) that prematurely discontinuate the study treatment
To compare mean changes in symptom severity on the Clinical Global Impression Scale, Severity | 6 weeks.
  To compare changes in symptom severity on the Clinical Global Impression scale (Severity) between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4). A higher score on CGI-S means worse symptom severity. Minimum score: 1, maximum score: 7
To compare mean changes in symptom severity on the Clinical Global Impression Scale, Improvement | 6 weeks.
  To compare changes in improvement on the Clinical Global Impression scale (Improvement) between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4). A higher score on CGI-I means more improvement. Minimum score: 1, maximum score: 7
To compare the reasons for premature treatment discontinuation (EIPT vs. TAU) (stopping before visit 4 while started medication at visit 2 | 6 weeks.
  To compare the difference in reasons for premature treatment discontinuation between the treatment arms over the treatment period.
To compare changes in suicidal ideation between treatment arms. | 6 weeks.
  Changes on the Columbia-Suicide Severity Rating Scale (C-SSRS) throughout the study; EIPT vs TAU.Higher scores mean higer suicidal ideation (Scale 1) or suicidal behavior (scale 2). Minimum score: 0, maximum score per scale: 5.

CONTACTS AND LOCATIONS:
Locations (13):
- Medical University Innsbruck, Innsbruck, Austria
- Germany (6):
  - Bezirkskliniken Schwaben, Bezirkskrankenhaus Augsburg, Augsburg
  - Universitätsklinik für Psychiatrie und Psychotherapie Bielefeld, Bielefeld
  - LWL-Klinik Dortmund, Bereich Forschung & Wissenschaft, Dortmund
  - University Hospital Frankfurt am Main - Goethe University, Frankfurt am Main
  - Klinik für Psychiatrie und Psychotherapie der Universitätsmedizin Mainz, Mainz
  - Westfälische Wilhelms-Universität Münster, Münster
- Italy (4):
  - Universita degli Studi di Brescia, Brescia
  - University of Cagliari, Cagliari
  - Università degli studi della Campania Luigi Vanvitelli, Naples
  - Azienda Ospedaliero-Universitaria "Città della Salute e della Scienza di Torino", Turin
- Fundació Clínic per a la Recerca Biomèdica, Barcelona, Spain
- King's College London, Psychiatry & Cognitive Neuroscience, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR